CLINICAL TRIAL: NCT04686357
Title: Randomized Controlled Trial (RCT) Comparing Microbiome-driven Embryo Transfer (mET) by EMMA/ALICE Test vs Conventional Frozen Embryo Transfer (FET) of Blastocysts in Infertile Women at Their First IVF/ICSI Cycle
Brief Title: RCT to Assess the Impact of Microbiome Status in Infertile IVF Patients at Their First IVF/ICSI Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Reproductive & Genetic Hospital of CITIC-Xiangya (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUTH EMMA 1.0
Record Dates: First submitted 2020-12-18; First posted 2020-12-28 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-03

CONDITIONS: Infertility, Female; IVF
Keywords: Endometrial microbiota; microbiome treated embryo transfer; frozen embryo transfer; randomized clinical trial; endometrial microbiome metagenomic analysis; analysis of infectious chronic endometritis
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (mET) (Experimental): Microbiome-driven embryo transfer of a single vitrified blastocyst in an HRT cycle according to the EMMA/ALICE test results.
  Interventions: Diagnostic Test: EMMA/ALICE
- Control group (FET) (Active Comparator): Frozen embryo transfer of a single vitrified blastocyst in an HRT cycle according to the clinical standard practice.
  Interventions: Diagnostic Test: EMMA/ALICE

INTERVENTIONS:
Diagnostic Test: EMMA/ALICE — Before randomization, an endometrial biopsy (EB) sample will be collected from all participants between day 15 and 25 of a natural cycle or after around 120 hours of progesterone (P) impregnation during a standard HRT cycle. The results of the EMMA/ALICE test will be provided to participants and their gynecologists. Depending on the test results, there are 3 different possibilities:
  1. Normal result
  2. Ultralow or Dysbiotic result
  3. Abnormal result (pathogens) All probiotics and antibiotics that will be used in the study are already authorized by the local health authorities and will be prescribed under their technical data sheet/brochure conditions following the medical indications.
  Arms: Intervention group (mET)
Diagnostic Test: EMMA/ALICE — Before randomization, an endometrial biopsy (EB) sample will be collected from all participants between day 15 and 25 of a natural cycle or after around 120 hours of progesterone (P) impregnation during a standard HRT cycle. The results of the diagnosis will not be disclosed with the patients randomized into this arm nor with their gynecologists.
  Arms: Control group (FET)

SUMMARY:
Although the endometrium has been traditionally considered free of bacteria, recent studies have documented the presence of an endometrial microbiome. The uterine microbiome can be defined as Lactobacillus-dominated (<90% Lactobacillus spp.) or non-Lactobacillus-dominated (<90% Lactobacillus spp. with >10% of other bacteria). The presence of a pathogenic microbiota in endometrium was associated with significant decrease in implantation, pregnancy, ongoing pregnancy and live birth rates. Some of these pathogens microorganisms can also produce infection and inflammation that may lead to chronic endometritis.

Nowadays, the endometrial microbiome can be investigated with the EMMA test and the most known pathogens related with chronic endometritis can be detected with the ALICE test,both of them developed by Igenomix group. Our goal in this project is to investigate at what extent, if any, the analysis of the endometrial factor, at a microbiome level, in patients at their first IVF cycle improves their clinical outcome.

DETAILED DESCRIPTION:
Some authors have reported the existence of an endometrial microbiota present in healthy woman and different from that in the vagina. It is well known that the presence of pathogens (such as Gardnerella and Streptococcus) in the endometrium is related with infertility, pregnancy loss, premature rupture of membranes and preterm birth.

Another factor which has an impact on infertility is Chronic Endometritis (CE). It consists of a persistent inflammation of the endometrial mucosa and its prevalence in infertile patients has been estimated to be between 2.8 and 39%, although this percentage can reach up to 50 and 60% in patients with miscarriages and repeated implantation failure, respectively. The most common cause of CE is bacterial infection, but the traditional methods of diagnosis (histology, hysteroscopy and microbial culture) often give discordant results between them.

Based on all mentioned above, two molecular tests have been respectively developed by Igenomix (an international company that provides leading advanced services in reproductive genetics and infertility) to assess endometrial microbiome: EMMA (Endometrial Microbiome Metagenomic Analysis) and ALICE (Analysis of Infectious Chronic Endometritis). EMMA test analyses and quantifies all the bacteria present in the endometrium, showing the main bacterial genera present in significant amount in an endometrial sample; while ALICE test quantifies the amount of pathogens more often causing CE (Enterococcus spp., Enterobacteriaceae (Escherichia and Klebsiella), Streptococcus spp., Staphylococcus spp., Mycoplasma spp., and Ureaplasma spp.), Chlamydia and Neisseria, also in an endometrial sample.

The current project aims to investigate in a randomized way the potential improvement on the clinical outcome of Chinese infertile patients at their first IVF cycle considering a personalized diagnosis and treatment (when applicable) of their endometrial microbiome status with the EMMA/ALICE. To do that, only the outcomes of the first single embryo transfers performed after the inclusion of each patient will be considered.

Considering a 30% of possible drop-outs, a total of 1018 patients will be recruited (509 randomized in each group). They will be allocated on a balanced way (assigned by chance like the flip of a coin) in one of the two arms described below. Reproductive outcomes (defined following The International Glossary on Infertility and Fertility Care, 2017) will be compared between the two groups.

Data exported from the source documents will be duly codified and treated in order to protect the clinical and personal information of participants in accordance with the current local legislation.

All the statistical analysis performed on the data, as well as the procedures, will be registered in a detailed Statistical Analysis Plan (SAP) that will be developed during the study and before starting data analysis.

An interim analysis of this data is planned once 50% of the recruitment has been achieved. Besides and at that same moment, the study will be overseen by an independent Data Monitoring Committee.

All of the statistical procedures will be done systematically by both, intention to treat analysis (ITT) and per protocol analysis (PP). The ITT analysis will include all randomized patients recruited and assigned to one of the two groups after biopsy collection and before randomization. The PP analysis will be applied to those patients who adequately follow the protocol assigned according to their group and in whom the transfer of the good quality blastocyst is performed.

ELIGIBILITY:
* Inclusion criteria

  * Patients whose written IC approved by the EC has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
  * Patients undergoing their first IVF/ICSI cycle (first oocyte pick up, freezing all) with their own oocytes that will receive single embryo transfer of frozen blastocyst stage embryos (day 5/6) on an HRT cycle.
  * At least 2 morphologically good quality embryos already vitrified in blastocyst stage (day 5/6).
  * Maternal Age: ≤37 years to rule out embryo factor in aging patients.
  * BMI: 18.5 - 30.0 kg / m2 (both inclusive).
  * Normal ovarian reserve (defined as: AFC ≥ 8; AMH level ≥1.0 ng/ml and/or FSH < 8 mU/ml) before the controlled ovarian stimulation (COS) initiation.
  * Serum P levels ≤ 1.5 ng/ml, measured within 24 hours before the hCG administration in the COS cycle.
  * Negative serological tests for HIV, HBV, HCV, RPR.
* Exclusion criteria

  * Patients with repeated miscarriages (> 2 previous biochemical pregnancies or > 2 spontaneous miscarriages).
  * Male partner with severe male factor (spermatozoa < 2 million/ml). Semen donor is allowed.
  * Patients who are intrauterine device (IUD) carriers in the last 3 months before sample collection.
  * Adenomyosis or any pathological finding affecting the endometrial cavity such as polyps/sub-mucosal myomas, intramural myomas > 4 cm, or hydrosalpinx must be previously operated at least 3 months before the endometrial samples are obtained.(Note: Patients are allowed to participate if the pathology is corrected before performing any study procedure).
  * Embryos analysed using preimplantation genetic testing for aneuploidies (PGT-A)
  * Women who have received antibiotics in the last month previous to sample collection, except for the prophylaxis for the oocyte retrieval. In the control group, antibiotics cannot be provided during the ET cycle
  * Illness or unstable medical condition that may put at risk the patient's safety and her compliance in the study

Max Age: 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1018 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | From date of embryo transfer until 40 weeks
  The number of deliveries that resulted in at least one live birth per ET (transferred patient). Live birth is defined as the complete expulsion or extraction from a woman of a product of conception after 22 weeks of gestation, which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.

SECONDARY OUTCOMES:
Implantation rate | From date of embryo transfer until 5-6 weeks
  The number of gestational sacs observed by vaginal ultrasound at the 5th gestational week divided by the number of embryos transferred.
Clinical miscarriage rate | From date of embryo transfer until 20 weeks
  Number of spontaneous pregnancy losses in which a gestational sac/s was previously observed, per number of pregnancies.
Biochemical pregnancy rate | From date of embryo transfer until 5-6 weeks
  Number of pregnancies diagnosed only by βhCG detection without a gestational sac visualized by vaginal ultrasound at the 5th week of pregnancy, per number of pregnancies.
Ectopic pregnancy rate | From date of embryo transfer until 8 weeks
  Number of pregnancies outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Pregnancy rate | From date of embryo transfer until 2 weeks
  Pregnancy rate is the number of patients with positive serum level of beta-HCG per embryo transfer.
Obstetric complications | From date of embryo transfer until 40 weeks
  Type and number of obstetric complications during pregnancy
Delivery complications | From date of embryo transfer until 40 weeks
  Type and number of delivery complications
Cost-effectiveness between mET and FET groups | 30 months
  To estimate the average cost per patient in each treatment to achieve a live newborn.
Proportion of microorganism in the infertile study population | From date of EB collection until 3 months
  Relative abundance of each microorganism identified in EB samples

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Principal Investigator — Peking university Third Hospital, Beijing; QingXue Zhang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Fei Gong, Principal Investigator — Reproductive & Genetic Hospital of CITIC-Xiangya